# Carotid Revascularization and Medical Management for Asymptomatic Carotid Stenosis Trial

NCT02089217

9/24/2014



# 1. General Information About This Research Study

**Study Title: CREST-2** 

Name of Principal Investigator on this Study: Thomas G. Brott, M.D.

#### A. Study Eligibility and Purpose

You are being asked to take part in this research study because you have carotid artery disease with no symptoms. This is called asymptomatic carotid artery disease. Your carotid artery disease is caused by a thickened area (plaque) in your artery. The thickened area narrows the artery and may limit blood flow to your brain.

Participants in this study will receive either intensive medical management alone or intensive medical management and a surgical procedure to open the carotid artery. The main purpose of the study is to find out if medical management alone results in different rates of death or stroke than medical management and a surgical procedure.

As you read this form describing the study, ask any questions you have. Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you decide. Your participation is voluntary. You may decide not to participate and you may stop participating at any time during the study. If so, none of your current benefits or normal health care will be affected in any way. When you feel comfortable that all your questions have been answered, and you wish to take part in this study, sign this form in order to begin your participation. Your signature means you have been told about the study and the risks. Your signature on this form also means that you want to take part in this study.

#### **B.** Number of Participants

Overall, there will be about 2,480 people enrolled in this study across North America.

#### C. Additional Information You Should Know

The National Institute of Neurological Disorders and Stroke (NINDS), a branch of the US National Institutes of Health (NIH) is funding the study. The NINDS will pay your study doctor or the institution to cover costs related to running the study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

#### **Conflict of Interest**

Your doctor may be referring you to this study and if your doctor is also an Investigator in this study, he or she has a potential conflict by having two sets of interests (your well-being, and the scientific conduct of the study). If you are uncomfortable with your doctor working with you as part of this research study, but still wish to participate in the research, you may request to work with a different member of the research team.



# 2. What Will Happen To You While You Are In This Research Study?

The study team will describe the treatment options for carotid disease. The options include intensive medical management with or without opening the artery.

Intensive medical management includes treatments for lifestyle risk factors such as high blood pressure, high cholesterol, diabetes, and smoking cessation.

The options for opening the carotid artery include carotid endarterectomy (CEA) or carotid artery stenting (CAS).

CEA is surgical procedure. During CEA the thickened area (plaque) of the artery is removed through an incision (surgical cut) in the neck.

CAS consists of placing a metal device called a stent in the narrowed part of the artery to hold it open.

The study team will discuss the benefits and risks of each treatment with you.

You and your treating doctor will then decide whether CEA or CAS would be the best option to open your carotid artery.

After you have decided whether CEA or CAS is the best option for you, you will be put in one of the two following groups by chance (as in the flip of a coin):

- medical management alone
- medical management plus the procedure selected for opening the artery

You will have a 1 out of 2 chance of being in either group. Neither you nor your doctor will be able to choose which group you are placed into.

#### **Intensive Medical Management:**

All participants in the study will undergo intensive medical management.

You will have blood tests to evaluate your risk factors for a stroke.

You will take a regular strength aspirin tablet (325 mg) once a day.

You may take other medications to control various risk factors such as high blood pressure or high cholesterol.

The study doctor will also work with your primary care doctor on a program for weight loss, smoking cessation, exercise, and diabetes management, depending on your individual health needs.

You will also be enrolled in a risk factor management program called INTERVENT. This is a program that is used around the country and in other parts of the world that helps patients manage their risk factors.



Help in managing your risk factors will be done through telephone calls with one of the INTERVENT staff members. These staff members, or coaches, are healthcare workers who are not physicians. These coaches have been specially trained to follow the medical management plan your study doctors have recommended for you and help you figure out ways to follow them as completely as possible.

You will have 6 telephone conversations with your coach in the first 3 months of the program and then 1 every 3 months until you have been in the study for 1 year. After that you will have a telephone conversation with your coach every 6 months for the rest of the time you are in the study. Each call will last from 15-20 minutes. You will not have to pay anything for these telephone calls. Reports will be sent to your study doctor and study coordinator about how well you are doing in the program. Your study doctor or coordinator will talk with you about how you are doing and if you should change anything.

It is important that you participate in the INTERVENT coaching. Studies have shown that this coaching is very helpful to patients. Patients enrolled in the program had better results in controlling their risk factors than those who were not enrolled in the program. It is important that each participant in this study use the same program to manage their risk factors. Using the same program makes it more likely that the participants are working on their risk factors in a similar way. This allows for a more accurate evaluation of the results of this study by the study researchers after the study is completed.

# Follow-up assessments

You will have an in-person visit with a member of the study staff at 30-days after you have been randomized. You will have a follow-up visit at 4 months, 8 months, 12 months and then every six months thereafter for up to 4 years. At your 12-, 24-, 36-, and 48-month visit, you will have blood drawn to monitor your risk factors and the effectiveness of the medication you are taking. You will also have a test to measure your cholesterol levels at 30 days. If you are a diabetic, you will have a blood test every 6 months to measure how well your diabetes is being controlled. If your blood tests are not meeting treatment goals, your study doctor may have additional blood tests repeated. These blood tests are standard tests done in practice to monitor risk factors and you or your insurance will be billed for those tests. You will be asked questions about your health status and any changes in your health since your last visit.

An important part of this study is to see how treatment of your carotid artery disease might affect your thinking (cognition). Research staff at the University of Alabama at Birmingham will contact you by telephone to complete a 20-minute cognitive testing session. You will be called at baseline, 30 days and annually for the next 4 years. Patients whose primary language is not English will not take part in this testing.

You will also have a carotid duplex ultrasound performed at the 12-, 24-, 36-, and 48-month visit. A carotid duplex ultrasound is done using a probe that is placed against the outside of your neck, over the carotid artery. Sound waves from the probe produce an image of the blood flowing through the artery. It is possible that during follow-up, a small proportion of patients may develop a stroke. Under these circumstances, your carotid artery may be considered to be "symptomatic." The standard of care is to undergo either surgery or stenting to open the "symptomatic" carotid artery, and we will recommend the same approach for you. The final decision will remain with you and your treating physician. You



will continue medical management and we will continue to follow your progress as planned in the study.

#### If you will undergo **Carotid Endarterectomy (CEA)**:

The study doctor will review the entire procedure with you. You will sign a separate consent form for the CEA surgery. A general description of what will be done during the procedure is described below.

#### Before the CEA procedure

You will need to take aspirin in preparation for your procedure. This medication is intended to prevent your blood from clotting and will be prescribed by your doctor. You will also be started on medications for lowering cholesterol, blood sugar, and blood pressure as necessary and appropriate for you. You will have blood tests to evaluate your risk factors.

You will be given fluids and medicines to help you relax and keep you from feeling pain through a needle inserted into a vein. The procedure may be performed under general anesthesia (while you are asleep) or local anesthesia (medication injected into your neck like that used by dentists). Your doctor and anesthesiologist will decide which form of anesthesia is best for you.

#### During the CEA

Your doctor will make an incision in your neck to expose your carotid artery. Your doctor will give you additional blood thinning medication during the procedure to prevent blood clots from forming in the arteries. The doctor will then open up the artery and remove the plaque that is attached to the artery wall. The artery and then the incision will be sewn closed; a patch may be used, usually made of artificial material.

#### After the CEA

After your surgical procedure, you will take aspirin (325 mg tablet) daily indefinitely. In addition to this, your doctor may ask you to take other medications, such as medicine to control blood pressure, blood sugar, and cholesterol, as necessary for you. Your stroke risk factors will be managed as they are for the patients assigned to receive medical management alone.

#### Follow-up requirements after hospital discharge

As detailed above, you will need to return to visit your doctor for follow-up examinations at one month, 4 months, 8 months, 12 months and then every six months thereafter for up to 4 years or until the study is completed.

At the time of these visits, you will be asked about any symptoms you may have had and have your vital signs taken. You will be asked questions about your quality of life and physical capabilities. You will have a brief examination focusing on neurological function.



# If you will undergo **Carotid Artery Stenting (CAS)**:

The study doctor will review the entire procedure with you. You will sign a separate consent form for the CAS procedure. A general description of what will be done during the stenting procedure is described below.

#### Before the stent procedure

As early as forty-eight hours before the procedure, you will need to take aspirin and one other medication in preparation for your procedure. These medications are intended to prevent your blood from clotting and will be prescribed by your doctor. You will also be started on medications for lowering cholesterol, blood sugar, and blood pressure as necessary and appropriate for you. You will have blood tests to evaluate your risk factors. [The day of your procedure, an intravenous line will be started to give you fluids and medicines for sedation (to make you sleepy) and pain prevention.]

#### During the stent procedure

- Your surgeon will make a surgical cut in your groin after using some numbing medicine.
- A catheter (small plastic tube) will be placed through the cut into an artery in the groin.
- The catheter is carefully moved up to your neck to the blockage in your carotid artery.
- The surgeon will use moving x-ray pictures (fluoroscopy) to see the artery and guide the catheter to the correct position. Contrast material (x-ray dye) is also injected to obtain pictures of these arteries (angiogram). Care will be taken to use the least amount of x-ray and dye as is necessary to perform the procedure safely for you.
- The surgeon will give you additional blood thinning medication during the procedure to prevent blood clots from forming in the arteries.
- Procedures will be used to minimize the risk of debris (a plaque or other tissue that may break away from the artery walls during the stenting procedure) entering the artery. The surgeon may place an embolic protection device in your carotid artery. This device is used to capture debris.
- The narrowing in your carotid artery may first be enlarged with a balloon catheter, if needed.
- The stent will then be placed in the narrowed area. The stent is an elastic-like metal splint that has been placed onto a catheter, which is covered to hold it in place while it is being positioned in the carotid artery.
- After the stent is positioned across the part of your artery that is narrowed, it is released and allowed to expand on its own. Sometimes, a balloon may be needed to help expand the stent.
- When released, the stent enlarges the blood vessel at the point of narrowing. The catheter is then removed.
- If used, the embolic protection device will then be closed and removed, leaving only the stent in place.
- Over a period of three to four weeks, the inner lining of the artery will grow over the stent surface and the stent will become a permanent part of your artery.

#### After the stent procedure

You will be instructed to take medications for a period of four weeks (either clopidogrel 75 mg daily, or, if allergic to clopidogrel, ticlopidine 250 mg 1-2 tablets daily). You will also be required to take



aspirin 325 mg 1-2 tablets daily for the first 30 days, and aspirin 325 mg daily thereafter. A lower amount of aspirin may be substituted if you can not tolerate the higher dose of aspirin. For the first four weeks, the combination of the two medicines will help prevent blood clots from forming. After that, you will be instructed to continue taking aspirin every day indefinitely. In addition to these medications your physician may ask you to take other medications, such as medicine to control blood pressure, blood sugar, or cholesterol as necessary for you. Your stroke risk factors will be managed as they are for the patients assigned to receive medical management alone.

#### Follow-up requirements after hospital discharge:

You will need to return to visit your doctor for follow-up examinations at one month, 4 months, 8 months, 12 months and then every six months thereafter for up to 4 years or until the study is completed.

# 3. How Long Will You Be in This Research Study?

You will be in the study for up to four years.

# 4. Why You Might Want To Take Part In This Research Study

This study may not make your health better. However information learned in this trial will help to better care for patients with asymptomatic carotid disease in the future.

# 5. What Are the Risks Of This Research Study?

The risks of this study fall into three broad categories:

- 1. Risks of opening the artery. The main risks of opening the artery for CEA and CAS include stroke, heart attack, and death.
- 2. The risks of not opening the artery. The risk of not opening the artery is that patients might be at a higher risk of stroke than if they underwent opening the artery.
- 3. The risks of medical intervention. Medical intervention for risk factor control has risks associated with specific drug therapies.

#### Risks of Intensive Medical Intervention Drug Therapies

The only drug that is specifically required on this study is aspirin. All subjects in this study will take aspirin.

#### **Aspirin Side Effects**

Aspirin may cause side effects. Tell your doctor if any of these symptoms are severe or do not go away:

- nausea
- vomiting
- stomach pain
- heartburn



### Risks of Carotid endarterectomy (CEA)

The risks associated with the CEA procedure include:

- minor stroke (symptoms go away in 30 days) (occurs in less than 5% or 5 out of 100 patients)
- major stroke (occurs in less than 5% or 5 out of 100 patients)
- death (occurs in less than 1% or 1 out of 100 patients)
- long-term discomfort at the site of the surgical incision (occurs in less than 5% or 5 out of 100 patients)
- surgery may cause damage to the blood vessels resulting in bleeding or vessel narrowing. This may cause problems with neurological (nerve) function, depending on the severity. (occurs in less than 5% or 5 out of 100 patients)

Additional risks associated with carotid endarterectomy or anesthesia include

- temporary or permanent damage to nerves in your face
- lung infection
- heart attack
- kidney failure
- low blood pressure
- abnormal heart rhythms
- pulmonary embolism (a potentially life-threatening condition resulting from a blockage to an
  artery in the lungs which prevents the lungs from functioning properly). Wound complications
  including moderate bleeding and infection may occur in a small number of cases (less than 5%
  or 5 out of 100 patients).

#### Risks Carotid Artery stenting (CAS)

The stenting part of this trial may be considered investigational by the FDA. All of the stents and their components that will be used in this trial have been approved by the FDA and are commercially available. However, there is a chance that the devices may be used off-label depending on your level of stenosis and what combination of devices your surgeon feels is best for your care.

The risks associated with the stent procedure (which could use a carotid stent system with an embolic protection device) include:

- minor stroke (symptoms go away within 30 days) (occurs in less than 5% or 5 out of 100 patients)
- major stroke (occurs in less than 5% or 5 out of 100 patients)
- death (occurs in less than 5% or 5 out of 100 patients)



- pulmonary embolism (occurs in less than 1% or 1 out of 100 patients)
- bleeding (occurs in less than 1% or 1 out of 100 patients)
- infection (occurs in less than 1% or 1 out of 100 patients)
- blockage to the artery in the leg requiring surgical repair (occurs in less than 1% or 1 out of 100 patients)
- need for blood transfusion (occurs in less than 1% or 1 out of 100 patients)
- low blood pressure (occurs in less than 5% or 5 out of 100 patients)
- failure to deliver a stent to the treatment site(occurs in less than 1% or 1 out of 100 patients)
- migration of the stent (occurs in less than 1% or 1 out of 100 patients)
- carotid stent deformation (occurs in less than 1% or 1 out of 100 patients)
- carotid stent fracture or other damage to the stent (occurs in less than 1% or 1 out of 100 patients)
- abnormal heart rhythms (occurs in less than 5% or 5 out of 100 patients)

There may be discomfort or bleeding at the site of insertion of the catheter into the artery.

Risks that may be associated with the embolic protection device are:

- thrombosis (clot) of the filter (occurs in less than 1% or 1 out of 100 patients)
- filter entanglement on the stent or other damage to the stent (occurs in less than 1% or 1 out of 100 patients)
- mechanical failure of the device (occurs in less than 1% or 1 out of 100 patients)

On very rare instances, filter entanglement with the stent or failure to recover the filter could result in the filter coming off and remaining inside the vessel. In such a case, your doctor would use additional measures to remove the filter or stabilize it in the vessel so that it does not block blood flow. The enlarging of the carotid artery may cause damage to the blood vessels resulting in bleeding or vessel narrowing. This may cause problems with neurologic (nerve) function or death, depending on the severity.

There is a chance that the stent could be released before it reaches the part of your artery that is narrowed. It may be necessary to place another stent in the proper place. The presence of another stent with more stent material may increase the risk of blood clots forming.

The stent was designed to expand to fit the size of the artery; however, the rare possibility exists that the stent could move after it is placed. Depending on the location of the stent, your doctor may leave the stent where it is, or may perform another procedure to remove or replace it.



The stent is a foreign body. Although metals such as those used to make stents have been implanted for years in humans, including blood vessels of the heart, kidneys and legs, the long-term information regarding potential side effects when using these metals in the carotid artery is limited to 10-15 years.

Some research participants may be allergic to the contrast material (x-ray dye) or other medications used during the procedure. Occasionally contrast material or drugs may cause damage to other tissues or organs, especially kidney dysfunction or failure. Such damage could result in minor injury, serious injury or even death.

Stenting involves exposure to radiation through the use of fluoroscopy, an x-ray camera that allows real-time moving images of the arteries.

Subjects who undergo CAS will receive aspirin combined with clopidogrel or ticlopidine. Clopidogrel and ticlopidine are blood thinning medications routinely given to patients undergoing CAS to help the stent stay open. If you are already taking these medications, you will be asked to continue them. If you are not taking these medications, they will be started by your doctor with your CAS procedure.

Side effects of clopidogrel and ticlopidine

- Bleeding may occur in up to 1 out of 10 patients. Bleeding can be serious and sometimes lead to death.
- Thrombotic Thrombocytopenic Purpura (TTP): TTP is rare occurring in 1 in 250,000 people taking clopidogrel and 1 in 5,000 people taking ticlopidine. TTP is a blood clotting problem where blood clots form in blood vessels; and can happen anywhere in the body. TTP may cause death. Symptoms of TTP include:
- Purplish spots (called purpura) on the skin or in the mouth
- Yellowing of the skin or the whites of your eyes

#### Other risks

Patients who undergo CEA or CAS may receive a medication called a 'statin'.

Side effects of 'statin' medications

There are many 'statin' medications. Your doctor will choose one of these medications. Side effects are similar among commonly used 'statin' medications.

Common (occur in 1 out of 10 people)

- Nausea
- Sore throat
- Diarrhea

Rare (occur in less than 1 out of 100 people)

- Muscle pain or damage that could cause kidney damage
- Liver damage



#### **Blood draws**

The risks of drawing blood include pain, bruising, and rarely, infection at the site of the needle stick.

#### Narrowing of the treated artery

Even with a successful procedure, CEA or CAS, there is a chance that the treated area could become narrow again. This may require additional treatment, such as repeat angioplasty and/or surgery to reduce the chance of stroke that can be caused by the re-narrowing.

#### **Pregnancy and Birth Control:**

The study may involve unforeseeable risks to you or your fetus if you are pregnant. Therefore, pregnant women are excluded from this study. Should you become pregnant while taking part in this study, you must immediately notify your doctor.

- 1) Will women of child-bearing-potential be allowed to participate in this study? **Yes**: Women of child-bearing-potential will be able to participate in this study if they have a negative pregnancy test and agree to use acceptable birth control (see #5) since the risks to an unborn child are either unknown or potentially serious.
- Will pregnant and/or nursing women be allowed to participate in this study?
   No: There is not enough medical information to know what the risks might be to an unborn child carried by a woman who takes part in this study.
- 3) Do you need to have a pregnancy test done to be part of the study?No: A pregnancy test will be done as part of your normal clinical care and not part of the study.
- 4) Will men who are able to father a child be allowed to participate in this study? **Yes:** Men who are able to father a child are allowed to take part in this study.
- 5) What types of birth control are acceptable?
  Surgical sterilization
  Approved hormonal contraceptives (such as birth control pills, Depo-Provera)
  Barrier methods (such as a condom or diaphragm) used with a spermicide
  An intrauterine device (IUD)

#### Risk summary

- Many side effects go away shortly after the medication or surgical procedure is stopped, but in some cases side effects can be serious, long lasting, or may never go away.
- Some side effects may not be known.
- Side effects may range from mild to life-threatening. There may be a risk of death.
- Other drugs may be given to make side effects less serious and less uncomfortable.
- Talk to the researcher and/or your healthcare provider about side effects and ask any other questions.



## 6. What Other Choices Do You Have If You Don't Take Part In This Research Study?

You do not have to be in this study to receive treatment for your condition. Your other choices may include other procedures or medications which will be discussed by the physician with you. You should talk to the researcher and your regular physician about each of your treatment options before you decide if you will take part in this study.

# 7. Are There Reasons You Might Leave This Research Study Early?

Taking part in this research study is voluntary. You may decide to stop at any time. You should tell the researcher if you decide to stop and you will be advised whether any additional tests may need to be done for your safety.

In addition, the researchers may stop you from taking part in this study at any time:

- o if it is in your best clinical interest,
- o if you do not follow the study procedures,
- o if the study is stopped.

### 8. Will You Need To Pay For Any Of The Tests And Procedures?

You and/or your health plan will need to pay for all tests and procedures that are part of this study, including CEA or CAS, and the blood tests to monitor your risk factors because they are part of regular medical care for patients with carotid artery disease. If your insurance does not cover the costs of the blood pressure and cholesterol medications required by this study to control your vascular risk factors, then the study will provide these medications at no additional cost to you.

The INTERVENT lifestyle program will be provided to you by the study free of charge whether you have health insurance or not.

# 9. Will You Be Paid For Participating In This Research Study?

You will not be paid for taking part in this study.

# 10. What Happens If You Are Injured Or Become Ill Because You Were In This Research Study?

If you have side effects from the study treatment, you need to report them to the researcher and your regular physician, and you will be treated as needed. Your hospital will bill you or your insurer for these services at the usual charge. You or your health plan might also have to pay for other drugs or treatments which are given to help you control side effects. Mayo will not offer free medical care or payment for any bad side effects from taking part in this study.

Before you take part in this study, you should call your health insurer to find out if the cost of these tests and/or procedures will be paid for by the plan. Some health insurers will not pay for these costs. You will have to pay for any costs not covered by your health insurer.



If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the beginning of this form. Your hospital or physician's office will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

# 11. What Are Your Rights If You Are In This Research Study?

Taking part in this research study will not change your rights and benefits. Taking part in this research study does not give you any special privileges. If you decide to not participate in this study, or stop in the middle of the study, no benefits are taken away from you. You do not have to be in this research study to receive or continue to receive medical care.

You will be told of important new findings or any changes in the study or procedures that may affect you or your willingness to continue in the study.

# 12. What About Your Privacy?

We have obtained a **Certificate of Confidentiality** from the Department of Health and Human Services. The Certificate is designed to prevent us from being forced to disclose identifying information for use in any federal, state, or local civil, criminal, administrative, legislative, or other court proceeding, even if faced with a court subpoena. You should understand, however, that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. We may not withhold information if you give your insurer or employer or a law enforcement agency permission to receive information about your participation in this project. This means that you and your family must also actively protect your own privacy.

The Certificate does not prevent us from taking steps, including reporting to authorities, to prevent serious harm to yourself or others. Such disclosures will be made as described below.

#### The research team may share your information with:

- The Department of Health and Human Services (HHS), to complete federal responsibilities for audit or evaluation of this project;
- Public health agencies, to complete public health reporting requirements;
- Hospital or university representatives, to complete hospital or university responsibilities for oversight of this study; and
- Your primary care physician if a medical condition that needs urgent attention is discovered; Appropriate authorities to the extent necessary to prevent serious harm to yourself or others.

#### Authorization To Use And Disclose Protected Health Information

Your privacy is important to us, and we want to protect it as much as possible. By signing this form, you authorize this hospital and the investigators to use and disclose any information created or collected in the course of your participation in this research protocol. This information might be in



different places, including your original medical record, but we will only disclose information that is related to this research protocol for the purposes listed below.

This information will be given out for the proper monitoring of the study, checking the accuracy of study data, analyzing the study data, and other purposes necessary for the proper conduct and reporting of this study. If some of the information is reported in published medical journals or scientific discussions, it will be done in a way that does not directly identify you.

This information may be given to other researchers in this study, including those at other institutions, the study sponsor, representatives of the companies who manufacture the carotid stent systems, including representatives in the USA or other countries, or private, state or federal government parties or regulatory authorities in the USA and other countries responsible for overseeing this research. These may include the Food and Drug Administration, the Office for Human Research Protections, or other offices within the Department of Health and Human Services, and the Institutional Review Board responsible for the review and reporting of this protocol, including the NIH StrokeNet Central Institutional Review Board at the University of Cincinnati. Using your social security number or other information, data from this project may be linked with national or regional health-related databases to be used for research purposes only.

Often it is helpful for scientists to share information they get from studies in order to learn more about health and disease. Combining information from different studies may help scientists learn even more. This collection of information is called a database. Your study data may be sent to one or more databases, where it is will be stored with data from other studies. The databases may be kept at universities, government agencies or private companies. The data may include health information. Your name and any other identifying information will never be included in information that is sent to a database (this is called de-identification). Researchers will always have a duty to keep your information confidential.

#### **Information Disclosed to Study Sponsor**

If this information is given out to anyone outside of the study sponsor, the information may no longer be protected by federal privacy regulations and may be given out by the person or entity that receives the information. However, the sponsor will take steps to help other parties understand the need to keep this information confidential.

This authorization lasts until the end of the study. The study does not end until all data has been collected, checked (or audited) and analyzed. Sometimes this can be years after your study visits have ended. For example, this could happen if the results of the study are filed with a regulatory agency like the Food and Drug Administration.

If you stop authorization, the sponsor may continue to use your information already collected as part of this study, but will not collect any new information. Also, you will no longer be able to participate in the study.

If you sign this informed consent form, you are giving permission for the use and disclosure of your health information for purposes of this research study. You do not have to give this permission. Your



health care outside of the study, payment for your health care, and your health care benefits will not be affected if you choose not to sign this form. However, if you do not sign this form, you will not be able to participate in the study.

Your name and telephone number will be provided to the University of Alabama at Birmingham Survey Research Unit and the INTERVENT program to conduct the telephone assessments required as part of this study.

The researchers in this study would like to have your social security number on file. This number will be kept in a password-protected, encrypted database separate from the rest of the study data. The purpose of keeping participants social security numbers on file is to potentially link them in the future with national or regional health-related databases for research purposes only. The file containing any social security numbers will be destroyed at the end of the study.

| Please initia | al one of the following: |
|---|---|
| | I agree to allow the research staff to use my social security number only as described in this study. |
| | I do not wish to disclose my social security number. |
| 13. What | Will Happen to Your Samples? |
| No biologic | eal samples collected as part of this research study will be stored for future use. |

# 14. Who Can Answer Your Questions?

| You can call | At | If you have questions or concerns about |
|---|---|---|
| Principal Investigator:<br>Dr. Thomas Brott<br>Or | Phone:<br>904-953-2000 | Questions about the study tests and procedures |
| Dr. James Meschia | | Research-related injuries or emergencies |
| Study Coordinator:<br>(NAME) | insert SC's phone # | Any research-related concerns or complaints |
| University of<br>Cincinnati IRB | Phone:<br>513-558-5034 | Rights of a research subject |
| Research Subject<br>Advocate | Toll-Free:<br>800-889-1547 | Use of Protected Health<br>Information<br>or any research-related concerns<br>or complaints |

IRB #: 2014-4397



Approved: 9/24/2014
Do Not Use After: 9/23/2015

# 15. Summary and Enrollment Signatures

You have been asked to take part in a research study. The information about this study has been provided to you to inform you about this study.

- I have read the whole consent form, and all of my questions have been answered to my satisfaction.
- I am satisfied that I have been given enough information about the purpose, methods, risks, and possible benefits of the study to decide if I want to join.
- I know that joining the study is voluntary, and I agree to join the study.
- I know that I can call the investigator and research staff at any time with any questions or to tell them about side effects.
- I know that I may withdraw from the study at any time.
- A copy of this form will be put in my medical records and I will be given a copy of this completed form.

Please sign and date to show that you have read all of the above guidelines. Please do not sign unless you have read this entire consent form. If you do not want to sign, you don't have to, but if you don't you cannot participate in this research study.

| (Date / Time) | (Printed Name of Participant) |
|---------------|------------------------------------------------|
| | (Signature of Participant) |
| (Date / Time) | (Printed Name of Individual Obtaining Consent) |
| | (Signature of Individual Obtaining Consent) |